CLINICAL TRIAL: NCT02221206
Title: Clinical Observation for the Root Resorption With Mini-Screw Implant Anchorage-assisted Retraction of Maxillary Incisors
Brief Title: Volumetric Analysis of Root Resorption With Mini-Screw Implant Anchorage-assisted Retraction of Maxillary Incisors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Mengjie Wu, Associate Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSF81371167
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Dental Dysgnathia
Keywords: Mini-Screw implant anchorage; retraction of maxillary incisors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): mini-screw implant anchorage-assisted retraction of maxillary incisors
  Interventions: Device: Mini-Screw implant
- Control (No Intervention): regular maximum anchorage

INTERVENTIONS:
Device: Mini-Screw implant — Mini-screw implants (VectorTASTM8*1.4mm, Ormco Corporation, USA) were placed between maxillary first molar and second molar after local anesthetic on both sides
  Arms: Treatment

SUMMARY:
The intended study is designed as a prospective randomized controlled trial (RCT), comparing and contrasting the effect of mini-screw implant anchorage-assisted versus regular maximum anchorage by retracting the maxillary incisors.

DETAILED DESCRIPTION:
The objective of the clinical study proposal will be to investigate the performance of early root resorption in order to find out if the magnitude and direction of retraction is appropriate for the retraction of maxillary incisors following the mini-screw anchorage.

Therefore, the study will compare and contrast the efficacy and results of the volumetric measurement by CBCT.

Patients

Males or females whose diagnoses require implant anchorage treatment will be included in the study. Inclusion criteria for the study are as followings:

Orthodontic indication for skeletal anchorage Adequate bone quantity for a palatal implant in the CBCT Good oral hygiene and normal wound healing capacity

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic indication for skeletal anchorage
* Adequate bone quantity for a palatal implant in the CBCT
* Good oral hygiene and normal wound healing capacity

Exclusion Criteria:

* Patients with cheilognathopalatoschisis and other system syndromes associated with craniofacial anomalies
* Patients with immunodeficiency, diseases requiring a prolonged steroid usage, previous radiation therapy or chemotherapy
* Patients with metabolic bone diseases or uncontrolled endocrine disorders
* Alcohol or drug abuse
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Root resorption | 10 months after implant insertion
  orthodontic analysis was done by a Cone beam computed tomography (CBCT) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mengjie Wu, MD, DDS, Principal Investigator — Department of Orthodontics, Hospital of Stomatology, Zhejiang University
Locations (1):
- Department of Orthodontics, Hospital of Stomatology, Zhejiang University, Hangzhou, Zhejiang, China